CLINICAL TRIAL: NCT02613663
Title: Evaluation of Surgical Time, Post-operative Pain and Marginal Bone Loss in Immediate Implant Using "Nanobone" Versus "Autogenous Bone" for Treatment of Patients With Unrestorable Single Tooth: Randomized Controlled Trials.
Brief Title: Immediate Implant Using "Nanobone" Versus "Autogenous Bone" for Treatment of Patients With Unrestorable Single Tooth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Ahmed Nouby Adam, Samar Ahmed Nouby Adam, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAdam
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Immediate Implant With Bone Graft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immediate implants with nanobone graft (Experimental): Nano-hydroxyapatite bone graft fill the gap between immediate implant and labial bone wall.
  Interventions: Procedure: Immediate implants with nanobone graft
- immediate implants with autogenous bone graft (Active Comparator): Autogenous graft fill the gap between immediate implant and labial bone wall.
  Interventions: Procedure: immediate implants with autogenous bone graft

INTERVENTIONS:
Procedure: Immediate implants with nanobone graft — Extraction of unrestorable tooth replaced with immediate implant and use nanobone graft to fill the gap.
  Other Names: Nano-hydroxy apatite bone graft with immediate implants
  Arms: immediate implants with nanobone graft
Procedure: immediate implants with autogenous bone graft — Extraction of unrestorable tooth replaced with immediate implant and use autogenous bone graft to fill the gap.
  Other Names: autograft used with immediate implants.
  Arms: immediate implants with autogenous bone graft

SUMMARY:
A successful implant therapy require appropriate hard and soft tissue, perfect implant position, appropriate alveolar ridge architecture and integration of the implant. after tooth extraction bone resorption takes place and affect the quantity and quality of the bone resulting in inadequate bone volume for implant placement and future prosthetic restoration and impair the esthetic, so insertion of implant immediately following tooth extraction reduce bone loss and enhance esthetics.the fresh socket of extracted tooth is wider than the implant diameter and the distance between the implant and the bone called Peri-implant gap which influence the stability, osseointegration of the implants and esthetics. using bone graft in this gap between bone and implant enhance osseointegration and post-operative healing. autogenous bone graft considered the gold standard graft material for filling defects as it is osteogenic,osseoconductive and osseoinductive, however this approach obtained from the primary donor site for harvesting bone in the oral cavity which requires longer surgical procedure and produce not enough bone volume. there are several post-operative complication may happen as donor site morbidity and swelling,discomfort and pain, so alternative treatment has been suggested using biomaterials to fill the gap and reduce adverse effect of autogenous grafts.Several studies evaluate the success rate of implants with "autogenous" bone graft versus other synthetic guided bone regeneration materials. Nano porous grafting material as a new synthetic material "nanobone" nanocrystalline hydroxyapatite embedded in a porous silica gel matrix has oseoconductive and biomimetic properties integrate with the host bone. the sub-micron modification in bone substitutes enhance osteogenic property. the objective of this study is to measure surgical time, pain, implant stability and marginal bone loss in immediate implant placement with using autogenous bone graft versus nanobone graft.

DETAILED DESCRIPTION:
Immediate implant placement with Nanobone will offers great advantages for patients with unrestorable tooth as regards decrease surgical time, Post-Operative pain and marginal bone loss, increase implant stability compared to immediate implant with autogenous bone graft.Study is to be conducted in the oral medicine and periodontology department - Cairo University, Egypt. Post graduate clinic 1st floor old section. Unit Sirona2with LED light. Digital radiographic imaging will be carried out in the Oral Radiology Department, Faculty of Oral and Dental Medicine, Cairo University using digital intra-oral x-ray machine as well as CBCT imaging. Using CBCT determine the size and length of fixture will be used. After a traumatic extraction, using drills to prepare the socket for the implant. Standard drilling procedures are performed according to the manufacturer's instructions implant direct. The axis of the implant must correspond to the incisal edges of the adjacent teeth or be slightly palatal to this landmark. Place the exact size determined previously by CBCT. In the esthetic zone, the implant head should be a minimum of 3 mm apical to an imaginary line connecting the cemento-enamel junctions of the adjacent teeth and apical to the interproximal and crestal bone.The gap between the facial aspect of the implant and the buccal wall was filled with NanoBone.The flap will be scored and sutured in place without tension. While in the control group, Harvesting of the autogenous bone graft will be done. This group will be subjected to the same implant placement protocol as the study group. Postoperative care include; A dressing will be applied to the extraoral wound for 24 hours postoperatively in the control group, Patients will maintain on oral antibiotics (Amoxicillin/Clavulanic acid 1gm q12h) and analgesics (cataflam 50 mg q8h) for 5 more days. Chlorohexidine mouth wash will be prescribed for 2 more weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from unrestorable tooth that candidate for classical implant placement .
* Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.
* Good oral hygiene and teeth bounding the alveolar ridge is not periodontally affected.

Exclusion Criteria:

* Patients with any systemic disease that may affect normal healing.
* Patient with bad oral hygiene.
* Intra oral soft tissue defect that would affect the closure of the intra oral wound.
* Patients with severely atrophic ridges requiring a staged grafting procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Surgical time | during surgery
  device for measurement is stop watch, unit of measurement is minutes.
post-operative pain | during 3 days after surgery
  device for measurement is visual analog scale, unit of measurement is 1-10 scale.

SECONDARY OUTCOMES:
degree of implant stability | after 6 month from the surgery
  device of measurement is periotest, unit of measurement discrete number.
Marginal bone loss | after 6 month from the surgery
  device of measurement is digital radiograph, unit of measurement millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Samar Nouby, Principal Investigator — Oral and dental medicine faculty, Cairo university.
Locations (1):
- Faculty of Oral and Dental Medicine. Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chiapasco M. Early and immediate restoration and loading of implants in completely edentulous patients. Int J Oral Maxillofac Implants. 2004;19 Suppl:76-91. PMID 15635948
- [Result] Becker W, Becker BE. Flap designs for minimization of recession adjacent to maxillary anterior implant sites: a clinical study. Int J Oral Maxillofac Implants. 1996 Jan-Feb;11(1):46-54. PMID 8820122
- [Result] Costantino PD, Friedman CD. Synthetic bone graft substitutes. Otolaryngol Clin North Am. 1994 Oct;27(5):1037-74. PMID 7816433
- [Result] Nemeth Z, Suba Z, Hrabak K, Barabas J, Szabo G. [Autogenous bone versus beta-tricalcium phosphate graft alone for bilateral sinus elevations (2-3D CT, histologic and histomorphometric evaluations)]. Orv Hetil. 2002 Jun 23;143(25):1533-8. Hungarian. PMID 12577407
- See also: Rationale for the application of immediate load in implant dentistry: Part I. Implant Dentistry — http://www.ncbi.nlm.nih.gov/pubmed/15359155